CLINICAL TRIAL: NCT01089530
Title: Clinical Intervention Study in the Primary Care Setting of Patients With High Plasma Fibrinogen in Primary Prevention of Cardiovascular Disease
Brief Title: Clinical Intervention Study in the Primary Care Setting of Patients With High Plasma Fibrinogen (EFAP)
Acronym: EFAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: SCMFIC FAMILY DOCTORS CATALAN SOCIETY GRANT (Unknown)
Responsible Party: Jordi Gol i Gurina, IDIAP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P03/07
Record Dates: First submitted 2010-02-10; First posted 2010-03-18 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Cardiovascular Risk Factors
Keywords: Fibrinogen; Cholesterol; Cardiovascular risk factors; Primary prevention; High levels fibrinogen; High plasma fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Standard care (No Intervention)
  Interventions: Behavioral: Lifestyle intensive group

INTERVENTIONS:
Behavioral: Lifestyle intensive group — hipocaloric diet smoking cessation physical exercise

SUMMARY:
Objectives:

* To study the possible effects of an intensive lifestyle change program on, the plasma fibrinogen levels in patients with no cardiovascular disease, with a high fibrinogen and normal cholesterol levels, and moderate Cardiovascular Risk (CVR).
* To analyse whether or not the effect on fibrinogen is independent of the effect on lipids.

Methods: Controlled, randomised clinical trial in 13 Basic Health Areas (BHA) in L'Hospitalet de Llobregat (Barcelona) and Barcelona city. Of the 436 patients between 35 and 75 years with no cardiovascular disease, with a high plasma fibrinogen (> 300 mg/dl) and a plasma cholesterol < 250 mg/dl, 218 received a more frequent and intensive intervention, consisting of advice on lifestyle changes and treatment. The follow up frequency of the intervention group was every two months. The other 218 patients continued with their usual care in the BHAs. Fibrinogen, plasma cholesterol and other clinical biochemistry parameters were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 30 and 75 years, than in 2 analytical consecutive, separated by a minimum interval of 15 days, have fibrinogen plasma > 300 mg/dl and plasma Total cholesterol < 250 mg/dl.
* Acceptance through informed consent of the patient to participate in the study.

Exclusion Criteria:

* Patients receiving lipid lowering treatment (including dietary measures)
* Local or generalized, acute or chronic infection.
* Patients with a history of cardiovascular disease.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436
Dates: Start 2003-01; Study Completion 2006-12

PRIMARY OUTCOMES:
To evaluate the effect of an intensive intervention to modify lifestyle (hypocaloric diet, smoking cessation and physical exercise) in the fibrinogen levels. | 24 months

SECONDARY OUTCOMES:
To assess the effect of this intensive intervention in some modifiable cardiovascular risk factors. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- ABS Florida Sud, L'Hospitalet Del Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Rodriguez Cristobal JJ, Alonso-Villaverde Grote C, Trave Mercade P, Perez Santos JM, Pena Sendra E, Munoz Lloret A, Fernandez Perez C, Bleda Fernandez D; EFAP group. Randomised clinical trial of an intensive intervention in the primary care setting of patients with high plasma fibrinogen in the primary prevention of cardiovascular disease. BMC Res Notes. 2012 Mar 1;5:126. doi: 10.1186/1756-0500-5-126. PMID 22381072